CLINICAL TRIAL: NCT06095011
Title: Posture Correction for the Treatment of Cubital Tunnel Syndrome (CuTS)
Brief Title: Posture Correction in Cubital Tunnel Syndrome
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: pause in research for 6 mos
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000036074; 000 (Other: CTGTY)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be recruited through occupational hand therapy clinics throughout the Yale New Haven Hospital system
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- normal conservative management + posture training (Experimental): Participants will receive normal conservative management as well as posture training via the UpRight Go posture trainer. The device will be provided to participants with all supplies and instructions that come from the original manufacturer and will be walked through how to install and use the necessary smartphone application as well as wear the posture trainer. Participants will be asked to wear the device daily for six weeks with goals for the amount of time spent wearing the sensor each day provided by the smartphone app. Participants will return to clinic in six weeks to return the device and submit usage data, or will mail back the device. Devices will be cleaned with disinfectant wipes before use by future participants.
  Interventions: Device: UpRight Go
- normal conservative management only (standard of care) (No Intervention): Participants will receive conservative management.only: standard of care for initial treatment of cubital tunnel syndrome

INTERVENTIONS:
Device: UpRight Go — The UpRight Go posture trainer is a commercially available biofeedback sensor that externally attaches to the wearer via a necklace or silicon adhesive. It vibrates when it senses that the wearer is slouching and connects to a smartphone application which sets daily goals, tracks usage, and provides assistance and support. It complies with International Electrotechnical Commission (IEC) standards.
  Arms: normal conservative management + posture training

SUMMARY:
The primary objective of this study is to determine whether the UpRight Go posture trainer reduces the symptoms of cubital tunnel syndrome in patients who have not had corrective surgery, as determined by improvements in VAS scores for pain, numbness, and weakness.

DETAILED DESCRIPTION:
This is a randomized controlled, non-blinded trial. All patients who are eligible to participate and who consent to participate will be randomized to either receive standard of care treatment alone, or standard of care treatment with the additional intervention of posture training. The nature of the intervention prevents blinding. All patients will be followed for 6 weeks and evaluated for symptom improvement or resolution.

All patients aged 18 and older who present to clinic with cubital tunnel syndrome of any severity and who have not previously undergone surgical intervention for this condition will be eligible to participate in this study. All participants must be amenable to conservative management of CuTS, wearing a posture training device daily, completing the accompanying questionnaires throughout the study, and returning for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Adult patients, between 18 and 99 years old
* Exhibiting signs and symptoms consistent with cubital tunnel syndrome including but not limited to pain, numbness, or paresthesia in an ulnar distribution, loss of grip strength, or loss of fine motor control of the fingers.
* Nerve conduction study, electromyography, MRI or ultrasound results consistent with the diagnosis of cubital tunnel syndrome
* Ability to wear a posture trainer daily and manage the associated smartphone application and questionnaire

Exclusion Criteria:

* History of spinal surgery, hand surgery or hand/wrist fracture
* History of cubital tunnel release surgery or carpal tunnel syndrome
* Pregnancy or lactation
* Known allergic reactions to silicon
* Long-standing history of T2DM, documented neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain score for pain using a Visual Analogue Scale (VAS) | Baseline and 6 weeks
  Pain score assessed using a linear VAS: a straight horizontal line of fixed length (100mm) on which participants will mark the point on the line that they feel represents their perception of their current state. The VAS score is determined by measuring, in millimeters, from the left hand end of the line to the point that the patient marks. The scale ranges from "no pain" to "severe pain". The longer the distance on the line, the more pain.
Change in pain score for numbness using a Visual Analogue Scale (VAS) | Baseline and 6 weeks
  Pain score for numbness assessed using a linear VAS: a straight horizontal line of fixed length (100mm) on which participants will mark the point on the line that they feel represents their perception of their current state. The VAS score is determined by measuring, in millimeters, from the left hand end of the line to the point that the patient marks. The scale ranges from "no pain" to "severe pain". The longer the distance on the line, the more pain.
Change in pain score for weakness using a Visual Analogue Scale (VAS) | Baseline and 6 weeks
  Pain score for weakness assessed using a linear VAS: a straight horizontal line of fixed length (100mm) on which participants will mark the point on the line that they feel represents their perception of their current state. The VAS score is determined by measuring, in millimeters, from the left hand end of the line to the point that the patient marks. The scale ranges from "no pain" to "severe pain". The longer the distance on the line, the more pain.

SECONDARY OUTCOMES:
Change in The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | Baseline and 6 weeks
  The DASH questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. Each item is scored on a 5 point Likert scale. Total score ranges from 0 (no disability) to 100 (most severe disability). Higher scores indicate a greater level of disability and severity.
Change in strength testing via pinch/grip test | Baseline and 6 weeks
  Pinch testing involves the patient pinching a pinchmeter, which measures the strength of the patient's pinch. Grip testing involves the patient gripping a dynamometer. The force that the patient is able to exert on the pinchmeter/dynamometer is measured in lbs/kgs, Newtons, or Pascals, and a higher reading indicates a greater strength. This provides valuable information about how a patient's strength is affected by cubital tunnel syndrome.
Change in Medical Research Council (MRC) Scale for Muscle Strength | Baseline and 6 weeks
  The MRC Scale is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction). This score was defined as the sum of MRC scores from six muscles in the upper and lower limbs on both sides so that the score ranged from 60 (normal) to 0 (quadriplegic). The Criteria requires that each of the six muscle groups listed in the table are examined bilaterally.
Change in range of motion testing | Baseline and 6 weeks
  Patients will be asked to actively move their upper body through a series of movements and postures, testing for flexibility in the neck, shoulders, elbows, and wrists. Limitations in movement are recorded qualitatively, which indicates the potential presence of concomitant pathology in the upper extremities, which could affect a patient's response to treatment.
Change in two-point discrimination testing | Baseline and 6 weeks
  A caliper or two point discriminator is used to apply pressure to a patient's finger tips. The patient is then asked to determine if one or two points of pressure are present, with the distance between the two points changing. The lowest distance between two points that the patient can distinguish is recorded in millimeters. A smaller distance indicates better fine-touch sensation at the finger tips and can indicate the quality of sensory nerves at the distal upper extremity.
Change in Semmes-Weinstein monofilament testing. | Baseline and 6 weeks
  The Semmes-Weinstein monofilament (SWM) testing is one of the clinical tests that measures the response to a touching sensation of the monofilaments using a numerical quantity. The monofilament is a small strand of nylon attached to a plastic base at fixed spacing's from 2mm to 15mm. The provider uses this monofilament to check for loss of feeling on your foot.
Change in Boston Carpal Tunnel Syndrome (BCTS) questionnaire | Baseline and 6 weeks
  The BCTS is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. The Symptom Severity Scale (SSS) with 11 questions is scored on a Likert scale of 1-5 and the Functional Status Scale (FSS) with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as difficult. A final score is calculated for each scale (the sum of the individual scores divided by the number of items) and ranges from 1 to 5, with a higher score indicating a more severe handicap.
Hours per day device was worn | up to 6 weeks
  The mean hours per day device was worn
Time spent with good posture | up to 6 weeks
  The mean time spent with good posture while wearing the device

CONTACTS AND LOCATIONS:
Overall Officials: Elspeth Hill, MBChB, PhD, MRes, MRCS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No